CLINICAL TRIAL: NCT04486781
Title: A Phase II Trial of Pembrolizumab as Standard of Care + sEphB4-HSA in Chemotherapy Ineligible or Chemotherapy Refusing Patients With Metastatic Urothelial Carcinoma
Brief Title: A Study of Pembrolizumab+ sEphB4 in Metastatic Urothelial Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vasgene Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-001
Record Dates: First submitted 2020-07-08; First posted 2020-07-27 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Therapy (Experimental): All study participants will receive Pembrolizumab + sEphB4-HSA through a needle in a vein in their arm for an hour in an outpatient clinic. Pembrolizumab will be given at Day 1 of each 3 week cycle. The study drug (sEphB4-HSA) will be given at Day 1, 8, and 15 of each 3 week cycle.
  Interventions: Drug: Pembrolizumab + sEphB4-HSA

INTERVENTIONS:
Drug: Pembrolizumab + sEphB4-HSA — sEphB-HSA may prevent tumor cells from multiplying and blocks several compounds that promote the growth of blood vessels that bring nutrients to the tumor.

SUMMARY:
sEphB-HSA may prevent tumor cells from multiplying and blocks several compounds that promote the growth of blood vessels that bring nutrients to the tumor. The purpose of this study is to evaluate the combination of Pembrolizumab + sEphB4-HSA in the population of patients with previously untreated advanced (metastatic or recurrent) urothelial carcinoma who are chemotherapy ineligible or who refuse chemotherapy.

DETAILED DESCRIPTION:
The combination of Pembrolizumab + sEphB4-HSA will be given through an intravenous infusion (into a vein). Each cycle of sEphB4-HSA will be given at Day 1, 8, and 15 of each 3 week cycle. Each cycle of Pembrolizumab will be given at Day 1 of each 3 week cycle.

Participants may continue on study protocol as long as they continue to respond and remains clinically stable on study medication.

Patients may come off treatment for the following reasons:

* Disease progression.
* If tumor resolves.
* For participants who become pregnant.
* Incidence or severity of adverse drug reaction in this or other studies indicates a potential health hazard to subjects.
* Patient withdraws consent.
* Study termination by the Sponsor.
* Participants who are non-compliant with respect to taking drugs, keeping appointments, or having tests required for the evaluation of drug safety and efficacy.
* Participant's condition renders them unacceptable for further treatment in the judgment of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Age ≥ 18 years.
* Be treatment naïve and have advanced (metastatic or recurrent) pathologically proven urothelial carcinoma. Patients progressing more than 12 months of their last dose of platinum-based neoadjuvant or adjuvant chemotherapy are eligible.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function as defined in Table 1., all screening labs should be performed within 10 days of treatment initiation.
* Be ineligible for chemotherapy in the assessment of the treating physician or refusing chemotherapy in frontline setting. Cisplatin ineligibility is defined as Cresatinine Clearance (CrCl) < 60cc/min, NYHA class III hear failure, grade II neuropathy and grade II hearing loss, the latter two also apply to carboplatin-based chemotherapy.
* Be approved to begin treatment with pembrolizumab per standard of care and pembrolizumab must be available to the patient. Patient must enroll on this study prior to the receiving the second dose of pembrolizumab and prior to having restaging imaging after receiving pembrolizumab. Other PD1/PDL1 antibodies are now allowed.
* Have measurable disease based on RECIST 1.1. We request an OPTIONAL core biopsy from an accessible metastatic site after a minimum of 2 cycles of treatment AND prior to progression of disease to help the investigators better understand the activity of these drugs in tumor tissue.

In addition, we request an OPTIONAL collection of any surgical specimens obtained per standard of care during the study. For instance, specimens from metastasectomy while patient is undergoing therapy on this study.

Exclusion Criteria:

* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has a known history of active TB (Bacillus Tuberculosis)
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma potentially cured after surgery or prostate cancer that is under control by hormonal agents.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Treated brain metastases are allowed.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has New York Heart Association (NYHA) class 3 or 4, myocardial infarction, acute coronary syndrome, diabetes mellitus with ketoacidosis or chronic obstructive pulmonary disease (COPD) requiring hospitalization in the preceding 6 months; or any other intercurrent medical condition that contraindicates treatment with sEphB4HSA or pembrolizumab or places the patient at undue risk for treatment related complications.
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Uncontrolled hypertension is excluded- systolic blood pressure >140mmHg or diastolic >90mmHg. Patients experiencing white coat hypertension the office, may be considered eligible if blood pressure log at home is within acceptable limits AND upon review and agreement from the Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-08-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Estimate of the overall response rate (ORR) of the combination of Pembrolizumab + sEphB4-HSA in the patients with previously untreated advanced (metastatic or recurrent) urothelial carcinoma who are chemotherapy ineligible or who refuse chemotherapy | At study entry until completion (average of 60 months)
  Objective tumor response (OR), a derived endpoint, will be based responses as coded at each evaluation. A patient who experiences either a confirmed complete response (CR) or a confirmed partial response (PR) according to RECIST v1.1, will be classified as having experienced an objective response. To estimate the overall response rate (ORR) of the combination of Pembrolizumab + sEphB4-HSA in this population of patients, the number of patients who experience a confirmed complete response (CR) or a confirmed partial response (PR) will be divided by the number of eligible patients who began treatment.

SECONDARY OUTCOMES:
To estimate the progression free survival (PFS) in these patients | Day 1, 8, 15 (each 3 week cycle), 30 days after last dose (safety follow-up), every 6 weeks (follow-up), every 12 weeks (survival follow-up) (average of 60 months)
  Toxicity as assessed by CTCAE v5 will be documented in all eligible patients who begin treatment.
To estimate the overall survival (OS) in these patients | Baseline, Day 1, 8, 15 (each 3 week cycle), 30 days after last dose (safety follow-up), every 6 weeks (follow-up), every 12 weeks (survival follow-up) (average of 60 months)
  Overall survival (OS) is calculated as the time from start of protocol treatment until death from any cause. Patients who are alive at the time of analysis will be censored at the last date that they were documented alive. OS will summarized for all eligible patients who begin treatment.
To determine the tolerbility of the combination of Pembrolizumab + sEphB4-HSA in patients with previously untreated advanced urothelial carcinoma is more effective than the single agent pembrolizumab. | Day 1, 8, and 15 of each 3 week cycle
  Progression-free survival (PFS) is calculated as the time from start of protocol treatment until documentation of disease progression (as defined by RECIST v1.1) or until death from any cause, whichever comes first. Patients who are alive and have not progressed at the time of analysis will be censored at the last date that they were documented alive and free of progression. In addition, patients who begin another treatment (i.e. other than Pembrolizumab or sEphB4-HSA alone) prior to progressing, will be censored at the time of the start of the other treatment for the primary analysis of this endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Sarmad Sadeghi, MD, Principal Investigator — University of Southern California
Locations (1):
- Sarcoma Oncology Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No